CLINICAL TRIAL: NCT00297596
Title: A Phase II Trial of Trastuzumab and Oxaliplatin in Patients With Metastatic Breast Cancer
Brief Title: Trastuzumab and Oxaliplatin in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 77
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Metastatic; HER2/neu+
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients with HER2 positive breast cancer received treatment with oxaliplatin 130 mg/m2 IV day 1 and trastuzumab 6 mg/kg (following 8 mg/kg loading dose during cycle 1). Cycles were repeated every 21 days.
  Interventions: Drug: Trastuzumab; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be administered as an 8 mg/kg loading dose by intravenous (IV) infusion over 90 minutes on day 1 of cycle 1. Subsequent doses will be administered as a 6 mg/kg IV dose over 30 minutes.
  Other Names: Herceptin
Drug: Oxaliplatin — Oxaliplatin will be administered at a dose of 130 mg/ m2 over 120 minutes on day 1 of each cycle, following standard antiemetic premedications. 21 day cycles.
  For the first cycle, trastuzumab will be administered before oxaliplatin; however for subsequent cycles, oxaliplatin will be infused prior to trastuzumab
  Other Names: Eloxatin

SUMMARY:
This is a phase II study of the combination of oxaliplatin and trastuzumab as first or second line therapy in patients with stage IV, metastatic breast cancer

DETAILED DESCRIPTION:
Eligible patients will receive a minimum of six cycles of combination therapy. If a patient is still responding to the oxaliplatin at 6 cycles, the oxaliplatin may be continued with the trastuzumab up to 10 cycles at the investigator's discretion. After discontinuing the oxaliplatin/trastuzumab combination, patients should continue with single agent trastuzumab until disease progression.

Trastuzumab will be administered as an 8 mg/kg loading dose by intravenous (IV) infusion over 90 minutes on day 1 of cycle 1. Subsequent doses will be administered as a 6 mg/kg IV dose over 30 minutes. Oxaliplatin will be administered at a dose of 130 mg/ m2 over 120 minutes on day 1 of each cycle, following standard antiemetic premedications. 21 day cycles.

For the first cycle, trastuzumab will be administered before oxaliplatin; however for subsequent cycles, oxaliplatin will be infused prior to trastuzumab

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 18 years of age
* Histologically confirmed breast cancer that is HER2/neu positive (3+ by IHC or FISH +) and evidence of metastatic disease. Tumor may be of any estrogen and progesterone receptor type
* Measurable disease by RECIST and an ECOG ≤ 2
* Patients with known evidence of brain metastases are eligible if they are asymptomatic and have completed all therapy (surgery, radiotherapy, and/or steroids)
* Baseline LVEF value within the institutional normal range
* Any number of prior hormonal therapy treatments in the adjuvant setting or for metastatic disease. A subject must have progressed on hormonal therapy and all hormonal therapy (including birth control pills) must be discontinued at study entry.
* Prior chemotherapy in the adjuvant setting and up to one prior chemotherapy regimen for metastatic disease is allowed.
* Patients may have received one prior trastuzumab/chemotherapy containing regimen or prior single agent trastuzumab.
* Prior radiation therapy in the adjuvant setting or for metastatic disease, provided it was not to the only site of evaluable disease.
* All prior chemotherapy, trastuzumab and radiation therapy should be completed > 2 weeks before enrollment.
* Patients receiving bisphosphonate therapy are eligible. However, if bisphosphonate were started within < 2 months prior to enrollment, the bone lesions will not be evaluated for response and the patient must have another site of metastatic disease that is either measurable or evaluable for response.
* Patients must have recovered from toxicities due to prior therapy.
* Lab values in accordance with the protocol
* Patients must be nonpregnant and nonlactating. Patients of childbearing potential must implement an effective method of contraception during the study (birth control pills are not allowed).

Exclusion Criteria:

* Bone only disease are ineligible
* Patients who received more than 1 prior chemotherapy regimen for metastatic disease are ineligible.
* Patients with a history of other cancers except curatively-treated carcinoma of the cervix in situ or non-melanomatous skin cancer.
* Active serious infection or other underlying medical condition that would impair their ability to receive protocol treatment.
* Uncontrolled nervous system metastases
* Dementia or significantly altered mental status that would interfere with proper consenting.
* Receiving other investigational therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Yardley DA, Daniel D, Stipanov M, Drosick DR, Mainwaring M, Peyton J, Shastry M, Hainsworth JD. A phase II trial of oxaliplatin and trastuzumab in the treatment of HER2-positive metastatic breast cancer. Cancer Invest. 2010 Oct;28(8):865-71. doi: 10.3109/07357901003631031. PMID 20690802
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20690802

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxaliplatin/Trastuzumab: Patients with HER2 positive breast cancer received treatment with oxaliplatin 130 mg/m2 IV day 1 and trastuzumab 6 mg/kg (following 8 mg/kg loading dose during cycle 1). Cycles were repeated every 21 days. Oxaliplatin : Oxaliplatin will be administered at a dose of 130 mg/ m2 over 120 minutes on day 1 of each cycle, following standard antiemetic premedications. 21 day cycles. For the first cycle, trastuzumab will be administered before oxaliplatin; however for subsequent cycles, oxaliplatin will be infused prior to trastuzumab Trastuzumab : Trastuzumab will be administered as an 8 mg/kg loading dose by intravenous (IV) infusion over 90 minutes on day 1 of cycle 1. Subsequent doses will be administered as a 6 mg/kg IV dose over 30 minutes.
Period: Overall Study
Arm/Group | Oxaliplatin/Trastuzumab
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin/Trastuzumab
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 59 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Trastuzumab
Number analyzed (Participants) | 25
percentage of participants | 20 [4.3 to 35.7]

2. Secondary Outcome: Time to Progression
Description: Time-to-progression was defined as the interval from first study treatment until the date that breast cancer progression was documented, other treatment was given, or death occurred.
Time Frame: 18 months
Measure: Median (Full Range); unit: months
Arm/Group | Oxaliplatin/Trastuzumab
Number analyzed (Participants) | 25
months | 1.7 [0.5 to 12.3]

ADVERSE EVENTS:
Arm/Group | Oxaliplatin/Trastuzumab
Serious Adverse Events (participants affected / at risk) | 7/25
Other Adverse Events (participants affected / at risk) | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin/Trastuzumab (N=25)
Perforated appendix (Gastrointestinal disorders) | 1 (1)
Respiratory failure secondary to metastatic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Right lower lobe pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pathologic fracture of let proximal humeral diaphysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathologic fracture of right proximal humeral diaphysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Massive pleural effusion with total collapse of right lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin/Trastuzumab (N=25)
Nausea (Gastrointestinal disorders) | 13 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Fatigue (General disorders) | 20 (62)
Diarrhea (Gastrointestinal disorders) | 15 (38)
Allergic Reaction (General disorders) | 2 (3) — Hypersensitivity Reaction
Neuropathy - Sensory (Nervous system disorders) | 17 (52)
Vomiting (Gastrointestinal disorders) | 5 (9)
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Taste Alteration (Gastrointestinal disorders) | 2 (3)
Anorexia (Gastrointestinal disorders) | 7 (10)
Constipation (Gastrointestinal disorders) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Dehydration (Gastrointestinal disorders) | 2 (2)
Mood Alteration - Depression (Nervous system disorders) | 2 (5)
Heartburn/dypepsia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Fever (General disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 18 (48)
Hot flashes/flushes (Endocrine disorders) | 2 (4)
Insomnia (General disorders) | 4 (8)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 12 (34)
Neuropathy - Motor (Nervous system disorders) | 2 (3)
Nail Changes (Skin and subcutaneous tissue disorders) | 2 (3)
Neutrophils/ granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (16)
Platelets (Blood and lymphatic system disorders) | 9 (21)
Pulmonary/Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 8 (14)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 8 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain (NOS) (General disorders) | 18 (42)
Pain (headache) (Nervous system disorders) | 2 (2)
Reflux (Gastrointestinal disorders) | 2 (4)
Weakness (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.